CLINICAL TRIAL: NCT02784509
Title: Translational Investigation of Growth and Everyday Routines in Kids (TIGER Kids)
Brief Title: Translational Investigation of Growth and Everyday Routines in Kids
Acronym: TIGER Kids
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amanda Staiano, PBRC Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2016-028; 3092-51000-04A (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Childhood Obesity
Keywords: Physical Activity; Sedentary Behavior; Cardiometabolic Risk Factors; Childhood and Adolescence
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — An aliquot of sample will be stored in case further tests are needed and if further consent is obtained from the subject.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the effect of severe obesity on physical activity, sedentary behavior and cardiometabolic risk factors during childhood and adolescence and whether these associations are modified by race. Additionally, the study will investigate the contributions of (total, regional, and depot-specific) fat accumulation on changes in physical activity, sedentary behavior, and cardiometabolic risk factors during childhood and adolescence.

DETAILED DESCRIPTION:
The proposed study will establish a prospective pediatric cohort to identify intervention targets based on the location, timing, barriers, and facilitators of current physical activity and sedentary behavior in a child's day. The project will be a prospective examination of 340 African American and White girls and boys aged 10 to 16 years, including 50% who are classified as severely obese. State-of-the-art technology will be used including accelerometry to quantify physical activity, magnetic resonance imaging to quantify fat accumulation, and geographic position system and ecological momentary assessment to identify environmental and socio-emotional barriers and facilitators. In further detail, this study will examine the following objectives:

Objective 1: Determine the effect of severe obesity on physical activity, sedentary behavior, and cardiometabolic risk factors during childhood and adolescence and whether these associations are modified by race.

Objective 2: Investigate the contribution of (total, regional, and depot-specific) fat accumulation on changes in physical activity, sedentary behavior, and cardiometabolic risk factors during childhood and adolescence.

Objective 3: Determine barriers and facilitators of physical activity that are related to obesity, including environmental and socio-emotional factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-16 years
* Body weight < 500 lbs.
* Ability to understand instructions and complete all study procedures

Exclusion Criteria:

* Pregnant
* On a restrictive diet due to illness
* Significant physical or mental disabilities that impede walking, wearing accelerometer or GPS, or responding to EMA.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study aims to identify and recruit 340 boys and girls aged 10 to 16 years. The sample will be screened on the telephone in attempt to achieve a comparable sex and race distribution. An oversample will be taken for severely obese youth so they comprise approximately 50% of the sample (with the other 50% being distributed among normal weight, overweight, and obese status).
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, PhD, Principal Investigator — PBRC Assistant Professor
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kracht CL, Beyl RA, Maher JP, Katzmarzyk PT, Staiano AE. Adolescents' sedentary time, affect, and contextual factors: An ecological momentary assessment study. Int J Behav Nutr Phys Act. 2021 Apr 15;18(1):53. doi: 10.1186/s12966-021-01121-y. PMID 33858416
- [Background] Kepper MM, Staiano AE, Katzmarzyk PT, Reis RS, Eyler AA, Griffith DM, Kendall ML, ElBanna B, Denstel KD, Broyles ST. Using mixed methods to understand women's parenting practices related to their child's outdoor play and physical activity among families living in diverse neighborhood environments. Health Place. 2020 Mar;62:102292. doi: 10.1016/j.healthplace.2020.102292. Epub 2020 Feb 5. PMID 32479369
- [Background] Kracht CL, Katzmarzyk PT, Staiano AE. Comparison of abdominal visceral adipose tissue measurements in adolescents between magnetic resonance imaging and dual-energy X-ray absorptiometry. Int J Obes (Lond). 2021 Jan;45(1):104-108. doi: 10.1038/s41366-020-0621-8. Epub 2020 Jun 4. PMID 32499526
- [Background] Kracht CL, Champagne CM, Hsia DS, Martin CK, Newton RL Jr, Katzmarzyk PT, Staiano AE. Association Between Meeting Physical Activity, Sleep, and Dietary Guidelines and Cardiometabolic Risk Factors and Adiposity in Adolescents. J Adolesc Health. 2020 Jun;66(6):733-739. doi: 10.1016/j.jadohealth.2019.12.011. Epub 2020 Jan 25. PMID 31987725
- [Background] Kepper MM, Staiano AE, Katzmarzyk PT, Reis RS, Eyler AA, Griffith DM, Kendall ML, ElBanna B, Denstel KD, Broyles ST. Neighborhood Influences on Women's Parenting Practices for Adolescents' Outdoor Play: A Qualitative Study. Int J Environ Res Public Health. 2019 Oct 12;16(20):3853. doi: 10.3390/ijerph16203853. PMID 31614711
- [Background] Kracht CL, Chaput JP, Martin CK, Champagne CM, Katzmarzyk PT, Staiano AE. Associations of Sleep with Food Cravings, Diet, and Obesity in Adolescence. Nutrients. 2019 Nov 30;11(12):2899. doi: 10.3390/nu11122899. PMID 31801259
- [Background] Kracht CL, Katzmarzyk PT, Champagne CM, Broyles ST, Hsia DS, Newton RL Jr, Staiano AE. Association between Sleep, Sedentary Time, Physical Activity, and Adiposity in Adolescents: A Prospective Observational Study. Med Sci Sports Exerc. 2023 Jan 1;55(1):110-118. doi: 10.1249/MSS.0000000000003018. Epub 2022 Aug 12. PMID 35977103
- [Background] Staiano AE, Katzmarzyk PT. Visceral, subcutaneous, and total fat mass accumulation in a prospective cohort of adolescents. Am J Clin Nutr. 2022 Sep 2;116(3):780-785. doi: 10.1093/ajcn/nqac129. PMID 35544287
- [Background] Fowler LA, Kracht CL, Denstel KD, Stewart TM, Staiano AE. Bullying experiences, body esteem, body dissatisfaction, and the moderating role of weight status among adolescents. J Adolesc. 2021 Aug;91:59-70. doi: 10.1016/j.adolescence.2021.07.006. Epub 2021 Jul 29. PMID 34333320
- [Background] Hu K, Button AM, Tate CM, Kracht CL, Champagne CM, Staiano AE. Adolescent Diet Quality, Cardiometabolic Risk, and Adiposity: A Prospective Cohort. J Nutr Educ Behav. 2023 Dec;55(12):851-860. doi: 10.1016/j.jneb.2023.10.003. Epub 2023 Oct 27. PMID 37897452
- [Background] Chen S, Kracht CL, Beyl RA, Staiano AE. Temporal Changes in Energy-Balance Behaviors and Home Factors in Adolescents with Normal Weight and Those with Overweight or Obesity. Int J Phys Act Health. 2023;2(2):5. doi: 10.18122/ijpah.020205.boisestate. PMID 37675056
- [Background] Denstel KD, Beyl RA, Danos DM, Kepper MM, Staiano AE, Theall KT, Tseng TS, Broyles ST. An examination of the relationships between the neighborhood social environment, adiposity, and cardiometabolic disease risk in adolescence: a cross-sectional study. BMC Public Health. 2023 Sep 1;23(1):1692. doi: 10.1186/s12889-023-16580-0. PMID 37658323
- [Background] Kracht CL, Pochana SS, Staiano AE. Associations Between Moderate to Vigorous Physical Activity, Sedentary Behavior, and Depressive Symptomatology in Adolescents: A Prospective Observational Cohort Study. J Phys Act Health. 2023 Feb 1;20(3):250-257. doi: 10.1123/jpah.2022-0345. Print 2023 Mar 1. PMID 36724791
- [Background] Kracht CL, Wilburn JG, Broyles ST, Katzmarzyk PT, Staiano AE. Association of Night-Time Screen-Viewing with Adolescents' Diet, Sleep, Weight Status, and Adiposity. Int J Environ Res Public Health. 2022 Jan 15;19(2):954. doi: 10.3390/ijerph19020954. PMID 35055781
- [Derived] Kepper MM, Staiano AE, Broyles ST. The Potential for Bias across GPS-Accelerometer Combined Wear Criteria among Adolescents. Int J Environ Res Public Health. 2022 May 13;19(10):5931. doi: 10.3390/ijerph19105931. PMID 35627467
- [Derived] Fearnbach SN, Johannsen NM, Martin CK, Katzmarzyk PT, Beyl RA, Hsia DS, Carmichael OT, Staiano AE. A Pilot Study of Cardiorespiratory Fitness, Adiposity, and Cardiometabolic Health in Youth With Overweight and Obesity. Pediatr Exerc Sci. 2020 Apr 25;32(3):124-131. doi: 10.1123/pes.2019-0192. PMID 32335525
- See also: Temporal Changes in Energy-Balance Behaviors and Home Factors in Adolescents with Normal Weight and Those with Overweight or Obesity — https://scholarworks.boisestate.edu/cgi/viewcontent.cgi?article=1083&context=ijpah
- See also: Associations Between Moderate to Vigorous Physical Activity, Sedentary Behavior, and Depressive Symptomatology in Adolescents: A Prospective Observational Cohort Study — https://labs.pbrc.edu/pediatric-obesity/documents/120.pdf
- See also: The Potential for Bias across GPS-Accelerometer Combined Wear Criteria among Adolescents — https://labs.pbrc.edu/pediatric-obesity/documents/ijerph-19-059311.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- TIGER Kids Sample: 342 boys and girls ages 10 to 16 years from every weight category (normal weight, overweight, and obese). Used state-of-the-art technology, including activity trackers and global positioning system (GPS) information, to track physical activity, imaging to measure body fat, and messages sent through a mobile phone app (called ecological momentary assessment) to identify what motivates or prevents kids from being physically active. Participants attended an orientation session at Pennington Biomedical to learn about the study, sign consent and receive their activity tracking tools. These tools were returned at clinic visit approximately 1 week later. Assessments include body measurements, blood pressure, surveys, blood draw, dietary recall and body composition. Participants will repeated the activity monitor tracking and a second clinic visit 2 years later.
Period: Overall Study
Arm/Group | TIGER Kids Sample
Started | 342
Completed | 256
Not Completed | 86

BASELINE CHARACTERISTICS:
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 256
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 95
  White | 147
  More than one race | 0
  Unknown or Not Reported | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective 1 Primary Outcome: Change in Minutes of Sedentary Behavior, Light Physical Activity, and Moderate-to-vigorous Physical Activity
Description: Physical activity and sedentary behavior will be measured by a triaxial accelerometer (Actigraph GT3X+, Actigraph of Ft. Walton Beach, FL). The participant will be instructed to wear the accelerometer on an elasticized belt, on the left mid-axillary line. The Actigraph is one of the most common accelerometers used for scientific purposes. Participants will be encouraged to wear the accelerometer 24-hours per day for at least 7-days (plus an initial familiarization day and the morning of the final day), including 2 weekend days. Participants will also complete a Lifestyle survey to collect information including diet and physical activity habits.
Time Frame: Baseline and Year 2
Population: 284/342 children had complete accelerometry data and were therefore included in analysis.
Measure: Mean (Standard Deviation); unit: Minutes measured from accelerometers
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 284
Minutes measured from accelerometers
  Sedentary Time | 21.4 (6.8)
  Light Physical Activitiy | 7.6 (5.7)
  Moderate-to-vigorous physical activity | 1.0 (2.3)

2. Primary Outcome: Objective 2 Primary Outcome: Relationship Between Total Fat Accumulation and Change in Sedentary Behavior - Visceral Adipose Tissue
Description: Body composition will be determined by DXA and MRI. With DXA, total body fat and trunk fat will be measured by whole-body DXA using a GE iDXA scanner (GE Medical Systems, Milwaukee, WI) to quantify total and regional body fat (including trunk fat). MRI - Visceral fat, i.e. visceral adipose tissue, will be measured by water-fat shifting MRI using the General Electric Discovery 750w 3.0 Tesla (GE Medical Systems, Milwaukee, WI). IDEAL-IQ imaging technique will be used to generate water-only, fat-only, in-phase, and out-of-phase echoes in a single acquisition with a 20-second breath-hold. Sedentary behavior will be measured by a a triaxial accelerometer as described in outcome 1. Participants will also complete a Lifestyle survey to collect information including physical activity habits.
Time Frame: Baseline and Year 2
Population: 251 children out of 342 had complete data and were therefore included in analysis.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 251
liters | .6 (.5)

3. Primary Outcome: Objective 2 Primary Outcome: Relationship Between Total Fat Accumulation and Change in Sedentary Behavior - Adiposity
Description: as for outcome 2
Time Frame: Baseline and Year 2
Population: 251 children out of 342 had complete data and were therefore included in analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 251
grams | 70.7 (30.2)

4. Primary Outcome: Objective 2 Primary Outcome: Relationship Between Total Fat Accumulation and Change in Sedentary Behavior - Body Fat (%)
Description: as for outcome 2
Time Frame: Baseline and Year 2
Population: 251 children out of 342 had complete data and were therefore included in analysis.
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 251
percentage of body fat | 34.2 (10.4)

5. Primary Outcome: Objective 2 Primary Outcome: Relationship Between Total Fat Accumulation and Change in Sedentary Behavior. - Waist Circumfrence
Description: as for outcome 2
Time Frame: Baseline and Year 2
Population: 251 children out of 342 had complete data and were therefore included in analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 251
cm | 78.4 (17.9)

6. Secondary Outcome: Objective 1 Secondary Analysis: Change in Daily Moderate to Vigorous Physical Activity (MVPA) Minutes Between Years.
Description: MVPA measured by a triaxial accelerometer (Actigraph GT3X+, Actigraph of Ft. Walton Beach, FL) as described in outcome 1. Participants will also complete a Lifestyle survey to collect information including physical activity habits.
Time Frame: Baseline and Year 2
Population: 323 participants had accelerometry data for Year 0 and 213 participants had accelerometry data for Year 2
Measure: Mean (Standard Deviation); unit: Minutes/day
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 323
Minutes/day
  Year 0 | 33.35 (19.40)
  Year 2 | 26.21 (16.67)

7. Secondary Outcome: Objective 1 Secondary Analysis: Change in Days/Week of Physical Activity Between Years.
Description: as for outcome 6
Time Frame: Baseline and Year 2
Population: 323/213 participants had accelerometry data in Year 0/Year 2
Measure: Mean (Standard Deviation); unit: Days/week
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 323
Days/week
  Year 0 | 7.03 (1.60)
  Year 2: number analyzed (Participants) | 213
  Year 2 | 6.17 (1.56)

8. Secondary Outcome: Objective 2 Secondary Analysis: Relationship Between Fat Mass Accumulation and Change in Physical Activity.
Description: Body composition will be determined by DXA and MRI. With DXA, total body fat and trunk fat will be measured by whole-body DXA using a GE iDXA scanner (GE Medical Systems, Milwaukee, WI) to quantify total and regional body fat (including trunk fat). MRI - Visceral fat, i.e. visceral adipose tissue, will be measured by water-fat shifting MRI using the General Electric Discovery 750w 3.0 Tesla (GE Medical Systems, Milwaukee, WI). IDEAL-IQ imaging technique will be used to generate water-only, fat-only, in-phase, and out-of-phase echoes in a single acquisition with a 20-second breath-hold. Physical Activity will be measured by a triaxial accelerometer as described in outcome 1. Participants will also complete a Lifestyle survey to collect information including physical activity habits.
Time Frame: Baseline and Year 2
Population: 217 children out of 342 hand complete data and were therefore included in the analysis
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | TIGER Kids Sample
Number analyzed (Participants) | 217
Kilograms
  Visceral adipose tissue | 0.5 (0.4)
  Subcutaneous adipose tissue | 5.0 (4.6)
  Total abdominal adipose tissue | 5.5 (5.0)
  Lean mass | 36.7 (10.3)
  Fat mass | 20.8 (13.9)

ADVERSE EVENTS:
Time Frame: 2 years 3 months
Arm/Group | TIGER Kids Sample
All-Cause Mortality (participants affected / at risk) | 0/342
Serious Adverse Events (participants affected / at risk) | 0/342
Other Adverse Events (participants affected / at risk) | 0/342

LIMITATIONS AND CAVEATS:
A limitation to assessing sedentary behavior, affect, & context is measuring them in real-time outside of the laboratory setting. Real-time assessment of these may better address complexities of daily life. Another limitation is that the current study does not have access to the CoreScan proprietary algorithm, which impedes algorithm-specific recommendations. Population level differences may provide insight to software developers & researchers on the systematic differences between techniques.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT02784509/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT02784509/ICF_001.pdf